CLINICAL TRIAL: NCT04889872
Title: The PROGRESS Trial: A Prospective, Randomized, Controlled Trial to Assess the Management of Moderate Aortic Stenosis by Clinical Surveillance or Transcatheter Aortic Valve Replacement
Brief Title: PROGRESS: Management of Moderate Aortic Stenosis by Clinical Surveillance or TAVR
Acronym: PROGRESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-01
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Aortic Stenosis, Calcific; Aortic Valve Stenosis
Keywords: Transcatheter aortic valve replacement (TAVR); SAPIEN 3; SAPIEN 3 Ultra; SAPIEN 3 Ultra RESILIA; Moderate aortic stenosis; Aortic stenosis; Transcatheter heart valve
MeSH Terms: conditions — Aortic Valve, Calcification of; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- TAVR (Experimental): Transcatheter Aortic Valve Replacement (TAVR)
  Interventions: Device: SAPIEN 3 / SAPIEN 3 Ultra / SAPIEN 3 Ultra RESILIA
- CS (No Intervention): Clinical Surveillance (CS)

INTERVENTIONS:
Device: SAPIEN 3 / SAPIEN 3 Ultra / SAPIEN 3 Ultra RESILIA — Patients will be implanted with a SAPIEN 3 / SAPIEN 3 Ultra / SAPIEN 3 Ultra RESILIA heart valve
  Arms: TAVR

SUMMARY:
This study objective is to establish the safety and effectiveness of the Edwards SAPIEN 3 / SAPIEN 3 Ultra / SAPIEN 3 Ultra RESILIA Transcatheter Heart Valve systems in subjects with moderate, calcific aortic stenosis.

Following completion of enrollment, subjects will be eligible for enrollment in the continued access phase of the trial.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, multicenter study. Subjects will be randomized to either transcatheter aortic valve replacement (TAVR) with the SAPIEN 3 / SAPIEN 3 Ultra /SAPIEN 3 Ultra RESILIA THV or Clinical Surveillance.

ELIGIBILITY:
Key Inclusion Criteria:

1. 65 years of age or older at time of randomization
2. Moderate aortic stenosis
3. Subject has symptoms or evidence of cardiac damage/dysfunction
4. The subject or subject's legal representative has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent.

Key Exclusion Criteria:

1. Native aortic annulus size unsuitable for the THV
2. Anatomical characteristics that would preclude safe transfemoral placement of the introducer sheath or safe passage of the delivery system
3. Aortic valve is unicuspid or non-calcified
4. Bicuspid aortic valve with an aneurysmal ascending aorta > 4.5 cm or severe raphe/leaflet calcification
5. Pre-existing mechanical or bioprosthetic aortic valve
6. Severe aortic regurgitation
7. Prior balloon aortic valvuloplasty to treat severe AS
8. LVEF < 20%
9. Left ventricular outflow tract calcification that would increase the risk of annular rupture or significant paravalvular leak post-TAVR
10. Cardiac imaging evidence of intracardiac mass, thrombus, or vegetation
11. Coronary or aortic valve anatomy that increases the risk of coronary artery obstruction post-TAVR

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2250 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2037-06 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | 2 years
  Non-hierarchical composite of death, and heart failure hospitalization or event
Primary Safety Endpoint | 30 days
  Non-hierarchical composite of death, stroke, life threatening or fatal bleeding, acute kidney injury stage 4, hospitalization due to device- or procedure-related complication, and valve dysfunction requiring reintervention

SECONDARY OUTCOMES:
Death, stroke, or heart failure hospitalization | 2 years
  The number of patients that had this event
Alive and Kansas City Cardiomyopathy Questionnaire (KCCQ) score improvement ≥10 points from baseline sustained through 2 years | 2 years
  The number of patients that met all these criteria
Heart failure hospitalization | 2 years
  The number of patients that had this event
Left ventricle (LV) mass index | 2 years
  Echocardiographic measurement of the size of the left ventricle
Diastolic dysfunction ≥ Grade 2 | 2 years
  Echocardiographic measurement of the stiffness of the left ventricle.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Généreux, MD, Principal Investigator — Morristown Medical Center, Morristown, NJ, USA; Jeroen J Bax, MD, PhD, Principal Investigator — Leiden University Medical Center, Leiden, The Netherlands; Raj Makkar, MD, Principal Investigator — Cedars-Sinai Medical Center, Los Angeles, CA, USA
Locations (80):
- United States (65):
  - Heart Center LLC, Huntsville, Huntsville, Alabama
  - Tucson Medical Center, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Huntington Hospital, Pasadena, California
  - Eisenhower Desert Cardiology Center, Rancho Mirage, California
  - Bay Area Structural Heart at Sutter Health, San Francisco, California
  - Kaiser San Francisco Medical Center, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Stanford Univeristy, Stanford, California
  - UC Health Medical Center of the Rockies, Loveland, Colorado
  - Yale Universtiy, New Haven, Connecticut
  - The Cardiac & Vascular Institute Research Foundation, Gainesville, Florida
  - Baptist Health Research Center, Jacksonville, Florida
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Emory University Atlanta, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Saint Alphonsus, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Alexian Brothers Hospital, Lisle, Illinois
  - Ascension Via Christi St. Francis, Wichita, Kansas
  - Louisiana State University, New Orleans, Louisiana
  - Ochsner Clinical Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital Boston, Boston, Massachusetts
  - Minneapolis Heart Institue, St. Paul's, Minneapolis, Minnesota
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - Saint Luke's Hospital of Kansas City Mid America, Kansas City, Missouri
  - St. Patrick Hospital, Missoula, Montana
  - Mary Hitchcock Memorial Hospital, Lebanon, New Hampshire
  - Atlantic Health System Hospital Corp - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - University of Buffalo Kaleida Health, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - NYU Langone Health, New York, New York
  - Columbia University Irving Medical Center/NYPH, New York, New York
  - Rochester General Hospital, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - Moses Cone Memorial Hospital, Greensboro, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Mount Carmel Health System, Columbus, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Kaiser Permanente Northwest, Clackamas, Oregon
  - Providence Heart & Vascular Institute Portland, Portland, Oregon
  - Legacy Emanuel Medical Center, Portland, Oregon
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Shadyside, Pittsburgh, Pennsylvania
  - Pinnacle Health Harrisburg, Wormleysburg, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Baptist Memorial Hospital Memphis, Germantown, Tennessee
  - Methodist Le Bonheur Healthcare, Germantown, Tennessee
  - Parkwest Medical Center, Knoxville, Tennessee
  - Saint Thomas Health, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Ascension Texas Cardiovascular, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - HCA Houston Healthcare Medical Center, Houston, Texas
  - The University of Texas Health Science Center, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Methodist Hospital of San Antonio, San Antonio, Texas
  - Kaiser Mid Atlantic, McLean, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington
- Australia (4):
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Health, Clayton, Victoria
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Hamiton Health Services, Hamilton, Onterio
- Japan (4):
  - Kokura Memorial Hospital, Fukuoka, Kyushu
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Sakakibara Heart Institute, Fuchū, Tokyo
  - Keio University Hospital, Shinjuku, Tokyo
- Netherlands (3):
  - AMC Amsterdam, Amsterdam, North Holland
  - Leiden Universitair Medisch Centrum, Leiden, South Holland
  - Erasmus Rotterdam, Rotterdam, South Holland
- Switzerland (2):
  - Hôpitaux Universitaire de Genève, Geneva
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No